CLINICAL TRIAL: NCT06871267
Title: Dietary Modification In Patients With Inflammatory Bowel Diseases And Its Impact In Gut Microbiome
Brief Title: Dietary Modification In Inflammatory Bowel Disease Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024321-13563
Record Dates: First submitted 2025-02-24; First posted 2025-03-11 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- General Healthy Diet Group (Active Comparator): Participants in this group will follow the quarter-quarter-half plate diet based on the Malaysian Healthy Plate guideline.
  Interventions: Behavioral: General Healthy Diet
- Crohn's Disease Exclusion Diet (CDED) Group (Experimental): Participants in this group will follow the Crohn's Disease Exclusion Diet (CDED), which consists of three phases with specific dietary restrictions.
  Interventions: Behavioral: Crohn's Disease Exclusion Diet (CDED)

INTERVENTIONS:
Behavioral: General Healthy Diet — Participants will follow the quarter-quarter-half plate diet as per the Malaysian Healthy Plate guideline.
  Arms: General Healthy Diet Group
Behavioral: Crohn's Disease Exclusion Diet (CDED) — Participants will follow the Crohn's Disease Exclusion Diet (CDED), which consists of three phases with specific dietary restrictions.
  Arms: Crohn's Disease Exclusion Diet (CDED) Group

SUMMARY:
This research project aimed to develop a culturally appropriate Asian Inflammatory Bowel Disease Diet for the Malaysian population, based on the Crohn's disease exclusion diet (CDED). The study will be conducted in inflammatory bowel disease patients in University Malaya Medical Centre, which are ulcerative colitis and Crohn's disease patients. The objectives of this study are to assess the impact of diet in clinical outcome and gut microbiota changes in patients with inflammatory bowel disease (IBD). The study duration spans 24 weeks, during which comprehensive follow-ups will be conducted at 0, 6, 12, and 24 weeks, respectively. At each follow-up session, participants will be requested to provide stool and blood samples for meticulous assessment of clinical and biochemical responses.

DETAILED DESCRIPTION:
Inflammatory bowel disease is a chronic gut inflammation due to immune system dysregulation. Although the exact causes remain unknown, patients' dietary habits were shown to affect the disease activity depending on the food exposure, either proinflammatory or anti-inflammatory food. This randomized-controlled trial (RCT) study aims to improve the modified CDED diet that is acceptable for the Malaysian population at Universiti Malaya Medical Centre. This study comprised of three parts: (Part 1: In-depth interview to measure the acceptance of the diet, Part 2: Implementation of the CDED diet, Part 3: Identification of change in gut microbiome post dietary intervention). The duration of the study is two years.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Crohn's disease according to established clinical, endoscopic, and histological criteria.
* Mild to moderate diseases (150 to 220 points).
* Written informed consent obtained.

Exclusion Criteria:

* Presence of stoma.
* Surgery within 6 months prior to randomization.
* Patient on exclusive enteral nutrition (EEN).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-09-10 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
To improve the Asian Inflammatory Bowel Disease diet. | 24 weeks
  Implementing improvised dietary guidance based on CDED is suitable for Asian settings to see patients' adherence (%) based on the diet adherence rating scale questionnaire.
Number of Participants Achieving Clinical Response at Week 12 | 12 weeks
  Clinical response will be assessed based on Crohn's Disease Activity Index (CDAI) score. An improvement of clinical response is defined as <150 CDAI score at week 12.

SECONDARY OUTCOMES:
Change in Fecal Calprotectin Concentration from Baseline to Post-Intervention | 12 weeks
  The effectiveness of the diet will be assessed by measuring fecal calprotectin concentration (mg/kg) at baseline and after the 12-week intervention.
Changes in Gut Microbiota Composition Over Time (Baseline, Week 6, Week 12, Week 24) | Baseline, Week 6, Week 12, Week 24
  The gut microbiota composition of participants will be assessed at Baseline, Week 6, Week 12, and Week 24 using 16S rRNA sequencing and shotgun metagenomics. Changes in microbiota composition will be evaluated based on relative abundance (%) of bacterial taxa at the genus/species level.
Differential Distribution of Gut Microbiota Between Control and Intervention Groups at Weeks 6, 12, and 24 | Week 6, Week 12, Week 24
  The gut microbiota composition of participants following the Crohn's Disease Exclusion Diet (CDED) will be compared to those following the General Healthy Diet at multiple time points (Week 6, Week 12, and Week 24). Between-group differences will be evaluated based on relative abundance (%) of bacterial taxa at the genus/species level.

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Malaya Medical Centre, Kuala Lumpur, Petaling Jaya, Malaysia

IPD SHARING:
Plan to Share IPD: No